CLINICAL TRIAL: NCT03427736
Title: Pharmacokinetics of Anesthetics and Analgesics in Children and Adolescent
Brief Title: Anesthetics and Analgesics in Children
Acronym: ANA01
Status: Recruiting | Type: Observational
Sponsor: Chi Dang Hornik (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Chi Dang Hornik, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00088893
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Pain
MeSH Terms: conditions — Pain | interventions — Ketorolac Tromethamine; Hydromorphone; Ketamine; Oxycodone; Morphine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Left over specimens will be de-identified and sent to the NICHD biorepository at the end of the study. These specimens may be made available to other researchers. Future unspecified tests conducted may include genetic testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug of Interest: Individuals receiving anesthetics or analgesics per standard of care
  Interventions: Drug: Ketorolac Tromethamine; Drug: Hydromorphone; Drug: Ketamine; Drug: Oxycodone; Drug: Morphine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — IV ketorolac will be given per standard of care, not prescribed for this study
  Other Names: Toradol
Drug: Hydromorphone — IV Hydromorphone will be given per standard of care, not prescribed for this study
  Other Names: Hydromorphone hydrochloride; Dilaudid
Drug: Ketamine — IV Ketamine will be given per standard of care, not prescribed for this study
  Other Names: Ketamine Hydrochloride
Drug: Oxycodone — PO Oxycodone(solution or tablet) will be given per standard of care, not prescribed for this study
  Other Names: Oxycodone Hydrochloride
Drug: Morphine — IV Morphine will be given per standard of care, not prescribed for this study
  Other Names: Morphine Sulfate

SUMMARY:
The purpose of this study is to characterize the pharmacokinetic (PK) and safety profile of anesthetics and analgesics in children and adolescents.

DETAILED DESCRIPTION:
This is a research study to find out what the side effects are of certain drugs that are commonly used for pain and to put people to sleep for surgery. The researchers also want to know how the drug is broken down in the body. Participants will be given these drugs as they are prescribed by their regular doctor. As part of the participant's standard of care, doctors will perform tests, ask questions, review medical information and measure vital signs (heart rate, blood pressure, etc). The researchers will collect information that doctors have already written in the medical records. The research study team will collect blood from participants at certain time points depending on when the participant was first given the drug (up to 5 samples over the course of 10 to 48 hours). Examples of current and upcoming anesthetics and analgesics include, but are not limited to: ketorolac (Toradol), ketamine (Ketalar), oxycodone (OxyContin), and morphine (Kadian, MS Contin).

ELIGIBILITY:
Inclusion Criteria:

1. 0 to <18 years of age at time of enrollment (must see applicable appendix for details as not all appendices enroll across the entire age range)
2. Parent and/or participant (if applicable) is able to understand the consent process and provides informed consent and HIPAA Authorization (if applicable)
3. Participant provides assent as required by the institutional review board (IRB) or research ethics board (REB)
4. Receiving one or more drugs of interest (DOI) per local standard of care
5. Meeting DOI-specific inclusion criteria (See Appendices)

Exclusion Criteria:

1. Known pregnancy
2. Extracorporeal life support (i.e., ECMO, dialysis, ventricular assist device)
3. Any condition which would make the participant, in the opinion of the investigator, unsuitable for the study

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 60 participants will be enrolled to each of the study drug of interests (DOI) cohorts. Participants who satisfy eligibility criteria and are receiving one or more DOIs per standard of care will be consented into the study and assigned to the corresponding DOI cohort. DOI cohort assignments will be at the discretion of the treating physician based on the DOIs that are administered per standard of care. Participants will be selected from a variety of centers including but not limited to trauma and intensive care units. Participants will not be randomized. Participants may count towards 1 or more DOIs within the same 90-day period.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Clearance (CL) or apparent oral clearance (CL/F) | up to 48 hours post dose
Volume of distribution (V) or apparent oral volume of distribution (V/F) | up to 48 hours post dose
Elimination rate constant (ke) | up to 48 hrs post dose
Half-life (t1/2) | up to 48 hrs post dose
Absorption rate constant (ka) | up to 48 hrs post dose
Area under the curve (AUC) | up to 48 hrs post dose
Maximum concentration (CMAX) | up to 48 hrs post dose
Time to achieve maximum concentration (TMAX) | up to 48 hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hornik, PharmD, Principal Investigator — Duke Clinical Research Institute
Locations (13):
- United States (11):
  - Lucile Packard Children's Hospital, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Ann and Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center of Texas, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
All data collected is uploaded into the National Institute of Health Data Repository (DASH) at the end of the study (de-identified).
Time Frame: Data will be uploaded to the repository within 2 years of study completion. It will be maintained in the repository indefinitely.
Access Criteria: In order to have access, researchers have to complete a Data access request. NICHD will review the request and either approve or deny it. IRB approval must be obtained by the researcher to access the data.
  https://dash.nichd.nih.gov/Resource/DataRequestChecklist
URL: https://dash.nichd.nih.gov/